CLINICAL TRIAL: NCT02116010
Title: Phase I/II Clinical Trial Randomized, Multicentric, Open Label, Standard of Care (Silver Sulfadiazine) Controlled Aiming at Assessing Tolerance and Efficacy of Local Bacteriophage Treatment of Wound Infections Due to E. Coli or P. Aeruginosa in Burned Patients Using Pherecydes Pharma Anti-Escherichia Coli and Anti-Pseudomonas Aeruginosa Bacteriophages GMP Produced Cocktails . This Project is a European Research & Development (R&D) Project Funded by the European Commission Under the 7th Framework Programme for Research and Development Involving 7 Clinical Sites in EU.
Brief Title: Evaluation of Phage Therapy for the Treatment of Escherichia Coli and Pseudomonas Aeruginosa Wound Infections in Burned Patients
Acronym: PHAGOBURN
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phaxiam Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHAGOBURN
Record Dates: First submitted 2014-04-01; First posted 2014-04-16 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Wound Infection
Keywords: Wound Infection in burned patient
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- E. coli, Standard of care : Silver Sulfadiazine (Active Comparator): Burn wounds infected by E. coli treated with Standard of care : Silver Sulfadiazine
  Interventions: Drug: Standard of care : Silver Sulfadiazine
- E. coli, Phages cocktail (Experimental): Burn wounds infected by E. coli treated with Pherecydes Pharma Phages cocktail
  Interventions: Drug: E. coli Phages cocktail
- P. aeruginosa, Standard of care : Silver Sulfadiazine (Active Comparator): Burn wounds infected with P. aeruginosa treated with Standard of care : Silver Sulfadiazine
  Interventions: Drug: Standard of care : Silver Sulfadiazine
- P. aeruginosa, Phages cocktail (Experimental): Burn wounds infected by P. aeruginosa treated treated with Pherecydes Pharma Phages cocktail
  Interventions: Drug: P. Aeruginosa, Phages cocktail

INTERVENTIONS:
Drug: E. coli Phages cocktail — Use of Pherecydes Pharma Phages cocktail to treat respectively E. coli burn wound infection
  Arms: E. coli, Phages cocktail
Drug: Standard of care : Silver Sulfadiazine — Use of Standard of care : Silver Sulfadiazine, to treat E. coli or P. aeruginosa infected burn wound
  Arms: E. coli, Standard of care : Silver Sulfadiazine; P. aeruginosa, Standard of care : Silver Sulfadiazine
Drug: P. Aeruginosa, Phages cocktail — Use of Pherecydes Pharma Phages cocktail to treat P. aeruginosa burn wound infection
  Arms: P. aeruginosa, Phages cocktail

SUMMARY:
The objective of PHAGOBURN is to assess tolerance and efficacy of local bacteriophage treatment of E. coli or P. aeruginosa wound infections in burned patients.

DETAILED DESCRIPTION:
PHAGOBURN is a Phase I/II clinical trial randomized, multicentric, open label, standard of care (Silver Sulfadiazine) controlled aiming at assessing tolerance and efficacy of local bacteriophage treatment of wound infections due to E. coli or P. aeruginosa in burned patients using Pherecydes Pharma anti-Escherichia coli and anti-Pseudomonas aeruginosa bacteriophage cocktails GMP produced. This project is a European Research & Development (R&D) project funded by the European Commission under the 7th Framework Programme for Research and Development. This project is involving 7 clinical sites in EU.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Adult Informed consent obtained from patient or next of kin
* In-hospital patient treated for burn wounds in a burn unit
* Burn wound (grafted or not) or graft harvesting area, presenting local signs of infection defined by SFETB criteria:

  * A local or loco-regional inflammatory reaction;
  * And/or an adverse and unexpected local evolution;
  * And/or regarding burn wounds: presence of pus, fast spontaneous debridement and separation, occurrence of blackish spots (necrosis or haemorrhage), unexplained conversion from a superficial lesion to a deep one (> 48th hour);
  * And/or regarding graft donor sites: presence of pus, unexplained delay in epidermisation, bedsore;
  * And/or regarding graft recipient sites: presence of pus, lysis of grafts, necrosis of fat located under the graft.
* Burn wounds with a microbiologically documented infection, as defined by positive surface swab, due to Escherichia coli or Pseudomonas aeruginosa whatever their resistance profile
* Treated by povidone-iodine

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Intercurrent condition requiring a treatment which may interfere with analysis results: such as high dose of chronic corticotherapy, immunosuppressive medication, oncologic chemotherapy
* Patient included in an interventional research protocol with therapeutic intervention still ongoing upon inclusion time or having participated into anti-infective drug trials during the previous month.
* Patient considered as part of a vulnerable population
* Patient for whom treatment limitation or withdrawal during study period is considered
* Allergy to Silver Sulfadiazine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Time for bacteria reduction adjusted on antibiotic treatment | 7 days
  Time necessary for a persistent bacteria reduction of two modes or persistent bacteria eradication relative to D0 adjusted on antibiotic treatment (active on targeted strain) introduced between D1 to D7. Bacteria count performed on bacteria targeted by the phages cocktail collected from surface swab samples assessed by the microbiologist.

SECONDARY OUTCOMES:
Assessment of tolerance of treatment | 21 days
  Adverse events frequencies will be assessed in each treatment arms. Phages therapy safety profile will be compared to safety profile of standard of care .
Incidence an delay of infection reduction with different bacterial species from the targets | 7 days
  The criteria will be assessed according to wound clinical examination and bacteria count by the microbiologist.
number of sites cured | 7 days
  The number of infected burns or infected wounds getting a clinical improvement will be described and compared between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Jault, MD, Principal Investigator — Service de Santé des Armées, Hopital Percy (Clamart, France)
Locations (5):
- Belgium (2):
  - Hopital Militaire Reine Astrid, Brussels
  - CHU Sart-Tilman, Liège
- France (2):
  - Hôpital d'instruction des armées Percy, Clamart
  - Centre hospitalier ST Joseph et St Luc, Lyon
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Derived] Jault P, Leclerc T, Jennes S, Pirnay JP, Que YA, Resch G, Rousseau AF, Ravat F, Carsin H, Le Floch R, Schaal JV, Soler C, Fevre C, Arnaud I, Bretaudeau L, Gabard J. Efficacy and tolerability of a cocktail of bacteriophages to treat burn wounds infected by Pseudomonas aeruginosa (PhagoBurn): a randomised, controlled, double-blind phase 1/2 trial. Lancet Infect Dis. 2019 Jan;19(1):35-45. doi: 10.1016/S1473-3099(18)30482-1. Epub 2018 Oct 3. PMID 30292481